CLINICAL TRIAL: NCT06312878
Title: CT Features of Interrupted Inferior Vena Cava With Azygous Continuation : a Retrospective Study
Brief Title: CT Features of Interrupted Inferior Vena Cava With Azygous Continuation
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN052024/CHUSTE
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Anatomical Variant of the Inferior Vena Cava
Keywords: Interrupted vena cava; Azygous continuation; Polysplenia; CT scan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included patients: All patients with interrupted IVC with azygous continuation on CT scan.
  Interventions: Other: Describe the anatomy of the IVC in the case of an anatomical variant

INTERVENTIONS:
Other: Describe the anatomy of the IVC in the case of an anatomical variant — Evaluated technique by collecting data from the medical record.

SUMMARY:
Inferior vena cava (IVC) is the largest vein is the body, draining blood from the abdomen, pelvis and lower extremities. IVC anomalies can be congenital or acquired.

The origins of these anomalies are not entirely clear, and their incidence is uncertain.

Imaging plays a pivotal role in diagnosis to prevent misinterpretation. CT scan is a quick, available, and suitable imaging modality in emergency setting.

The aim of this retrospective monocentric study was of describe CT features of interrupted suprarenal inferior vena cava with azygous continuation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with interrupted IVC with azygous continuation on CT scan were included in this study.

Exclusion Criteria:

* Patients under 18 years of age
* Patients no available CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with interrupted IVC with azygous continuation on CT scan
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Describe CT features of interrupted suprarenal inferior vena cava with azygous continuation | Day : 1
  The number of infrarenal inferior vena cava was recorded for each patient.

SECONDARY OUTCOMES:
Describe CT features of interrupted suprarenal inferior vena cava with azygous continuation | Day : 1
  The type of drainage of the left renal vein was recorded for each patient.
Describe association with polysplenic syndrome | Day : 1
  Measurement of splenic laterality
Describe association with polysplenic syndrome | Day : 1
  Measurement of stomach laterality
Describe association with polysplenic syndrome | Day : 1
  Measurement of liver morphology
Describe association with polysplenic syndrome | Day : 1
  Measurement of the preduodenal portal vein
Describe association with polysplenic syndrome | Day : 1
  Measurement of pancreatic and intestinal rotation malformations
Describe association with polysplenic syndrome | Day : 1
  Measurement of cardiopulmonary malformations
Describe circumstances of discovering the interrupted IVC | Day : 1
  The circumstances of discovering the interrupted IVC were also documented from clinical records.
Describe circumstances of discovering the interrupted IVC | Day : 1
  An history of thrombotic events was also documented from clinical records.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain GRANGE, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No